CLINICAL TRIAL: NCT05114200
Title: Evaluation of Drug Spread in Ultrasound-Guided Erector Spina Plane Block With Fluoroscopy
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Halil Cetingok, Assistant Professor, Istanbul University
Other Study IDs: 2021/467
Record Dates: First submitted 2021-09-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pain, Myofacial; Back Pain
Keywords: Erector spinae plane block
MeSH Terms: conditions — Facial Pain; Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: erector spinae plane block applied patients
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Patients will be placed in prone position. Mild sedation will be achieved by using 1-2 mg of midazolam and 50-75 µg of fentanyl iv. The application area will be visualized with General Electrics (GE) Logiq e Ultrasound device using 10-12 MHz linear probe or convex probe. Transverse process and erector spinae muscles will be visualised at the target vertebral level. Following local anesthesia (1-2 cc 2% lidocaine) application to the insertion site, a 20 gauge spinal needle will be inserted using the "in-plane" technique. The needle will be advanced up to the transverse process under ultrasound guidance. After confirming needle position with hydrodissection, 40 mg triamcinolone, 10 cc 0,5% bupivacaine, 10 cc radiopaque contrast agent solution will be injected. Imaging will performed in AP and lateral positions with fluoroscopy immediately and 30 minutes after the injection to evaluate intectate spread.

SUMMARY:
The purpose of this study is to evaluate the injectate spread in erector spinae plane blocks under fluoroscopy.

DETAILED DESCRIPTION:
The study will be carried out between March 2021 and June 2021 in Istanbul University Istanbul Medical Faculty Pain Medicine Clinic. Patients who undergone erector spinae plane block for any indication over the age of 18 will be included in the study.

All procedures will be performed in the operating room under standard monitorization (ECG, pulse oximetry, non-invasive blood pressure) and all patients will be in the prone position. The application area will be sterilized with povidone-iodine solution. Mild sedation will be achieved by using 1-2 mg of midazolam and 50-75 µg of fentanyl iv. The target area will be visualized by General Electrics (GE) Logiq e Ultrasound device using a 10-12 MHz linear probe or 1-4 MHz curvilinear probe. Transverse processes and erector spina muscles will be visualised at the target vertebral level. After local anesthesia (1-2 cc 2% lidocaine), a 20 gauge spinal needle will be inserted using the "in-plane technique". The needle will be advanced to the transverse process, after it's position is confirmed with hydrodissection, a solution of 40 mg triamcinolone, 10 ml 0,5% bupivacaine, 10 ml radiopaque contrast agent will be injected. Contrast spread will be evaluated with the fluoroscopy in the anterior-posterior and lateral positions immediately and 30 minutes after the procedure. The level of contrast radiating in the AP plane and passing through the paravertebral space and the epidural distance in the lateral plane will be noted. In addition, sensory examination with a pin prick test will be performed to determine the presence of dermatomal hypoalgesia and/or analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old
2. Patients who underwent erector spinae plane block for any reasons

Exclusion Criteria:

1. Age under the age of 18
2. Patients without a clear contrast spread under fluoroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent erector spinae plane block for any reasons
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The level of contrast spread in the anteroposterior plane | 0 minutes
  Fluoroscopic images will be taken in the anteroposterior plane, number of vertebral levels the injectate has spread out will be recorded.
The level of contrast spread in the anteroposterior plane | 30 minutes
  Fluoroscopic images will be taken in the anteroposterior plane, number of vertebral levels the injectate has spread out will be recorded.

SECONDARY OUTCOMES:
Contrast spread to paravertebral space | 0 minutes
  Fluoroscopic images will be taken in the anteroposterior and lateral plane, and contrast spread to the paravertebral space will be recorded.
Contrast spread to paravertebral space | 30 minutes
  Fluoroscopic images will be taken in the anteroposterior and lateral plane, and contrast spread to the paravertebral space will be recorded.
Contrast spread to epidural area | 0 minutes
  Fluoroscopic images will be taken in the anteroposterior and lateral planes, and contrast spread to the epidural area will be recorded.
Contrast spread to epidural area | 30 minutes
  Fluoroscopic images will be taken in the anteroposterior and lateral planes, and contrast spread to the epidural area will be recorded.
Pinprick test | 0 minutes
  Pinprick test will be performed to determine hypoalgesia and/or analgesia in relevant dermatomes
Pinprick test | 30 minutes
  Pinprick test will be performed to determine hypoalgesia and/or analgesia in relevant dermatomes

CONTACTS AND LOCATIONS:
Overall Officials: Halil Cetingok, Ass. Prof., Principal Investigator — Istanbul University Istanbul faculty of medicine department of pain medicine
Locations (1):
- Halil Cetingok, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No